CLINICAL TRIAL: NCT05330351
Title: Evaluation of Gastric Contents by Ultrasound in Pediatric Trauma Patients Undergoing General Anesthesia
Brief Title: Gastric Ultrasound in Pediatric Trauma Patients
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 21-019564
Record Dates: First submitted 2022-03-14; First posted 2022-04-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Trauma; Complications; Aspiration
Keywords: pediatric; trauma; gastric; ultrasound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Trauma Patients: Pediatric patients (<18 years old) who have suffered a traumatic event requiring surgical fixation within 48 hours prior to time to arrival in the operating room.
  Interventions: Diagnostic Test: Gastric Ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound — The investigators will compare gastric fluid volume as determined by ultrasound pre-induction vs. gastric volume aspirated via an orogastric tube post-intubation. The results will be stratified into low risk, moderate risk and high risk for aspiration based on ultrasound exam by an investigator off-line.

SUMMARY:
Gastric ultrasound has become increasingly utilized to examine volume and quality of gastric contents in the preoperative setting to guide anesthetic management and relay risk of aspiration in both adult and pediatric medicine. Gastric fluid volumes in trauma patients are thought to be elevated due to delayed gastric emptying in the setting of an over-attenuated sympathetic response to physical pain and stress, opioid analgesia, and other associated injuries (traumatic brain). However, there is a paucity of literature examining gastric fluid volumes (GFV), measured by gastric ultrasound, in the pediatric trauma population. The purpose of the study is to assess whether preoperative gastric ultrasound is an accurate method to identify pediatric trauma patients who have elevated GFV (>0.8mL/kg) and high-risk gastric contents (solids, complex liquids, in addition to large volumes).

DETAILED DESCRIPTION:
There is longstanding evidence that GFV are elevated in trauma patients for several physiologic reasons. This has been corroborated in both adult and pediatric studies, suggesting that trauma patients may be at higher risk for gastric aspiration compared to healthy controls, and that anesthetic management should reflect this elevated risk. This often implies tracheal intubation with or without a rapid sequence induction. However, performing rapid sequence induction to decrease aspiration risk increases the risk of desaturation, hypoxia, bradycardia, and hemodynamic instability, especially in small children who have reduced functional residual capacity and who are difficult to adequately preoxygenate. This has presented a question-mark for anesthesia providers caring for children with traumatic injuries, and variations in practice. Bricker and authors examined gastric fluid volumes by aspiration of gastric contents in 1989 in pediatric trauma patients, and found that nearly 50% had elevated gastric contents and were at risk for potential aspiration, though no aspiration events were captured. Likewise, Schurizek and authors looked a cohort of pediatric patients presenting for emergency surgery, which included trauma, and found the nearly 38% of children presenting to the OR who had adequately fasted had elevated gastric contents. A recent study using gastric ultrasound in children with proximal limb fractures found a similar rate of elevated gastric contents with 37% of children meeting criteria, and 24% of those showing evidence of solids/complex gastric fluid. Again, no aspiration events were captured. Thus, little is known to inform anesthesiologists about which risk factors contribute to high gastric volumes in pediatric trauma patients or how long these children may be considered at additional risk for aspiration. Aspiration is an extremely rare event, typically estimated between 1-5/10,000 anesthetics or 0.01%, and the sample size needed to power a study to capture reducing the risk of aspiration is not feasible. Thus, the investigators hope to characterize gastric contents/GFV using ultrasound in pediatric trauma patients presenting with a wide variety of traumatic injury and at varying times from injury (urgent/emergent surgery versus semi-urgent surgery), to identify potential risk factors and guide anesthetic management in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ages 0-17 years-old
* Patients suffering from a traumatic injury requiring urgent or emergent surgery.
* Inpatient or Same-Day Surgery

Exclusion Criteria:

* Children with altered or abnormal gastric physiology, ie, history of Nissen Fundoplication, history of short-gut syndrome, history of bariatric surgery/gastric sleeve, history of gastroparesis or functional dysmotility, etc.

Ages: 0 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: perioperative pediatric trauma patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric fluid volume (GFV) | GFV will be measured immediately prior to induction of general anesthesia within the operating room.
  GFV will be estimated via obtained gastric antral cross-sectional area (CSA), measured by ultrasound, and calculated using the formula: GSV= 0.0093 * CSA [mm2] - 0.96. This calculated GFV will be compared to aspirated gastric volumes.

SECONDARY OUTCOMES:
Airway management patterns | This data will be collected up to 1 year.
  We will also collect data on airway management patterns in pediatric trauma patients (rapid-sequence induction, laryngeal mask airway, etc).
Aspiration | This data will be collected up to 1 year.
  Number of patients with aspiration intraoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Elaina Lin, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hardman JG, O'Connor PJ. Predicting gastric contents following trauma: an evaluation of current practice. Eur J Anaesthesiol. 1999 Jun;16(6):404-9. doi: 10.1046/j.1365-2346.1999.00513.x. PMID 10434171
- [Background] Schurizek BA, Rybro L, Boggild-Madsen NB, Juhl B. Gastric volume and pH in children for emergency surgery. Acta Anaesthesiol Scand. 1986 Jul;30(5):404-8. doi: 10.1111/j.1399-6576.1986.tb02439.x. PMID 3766097
- [Background] Power I, Easton JC, Todd JG, Nimmo WS. Gastric emptying after head injury. Anaesthesia. 1989 Jul;44(7):563-6. doi: 10.1111/j.1365-2044.1989.tb11442.x. PMID 2774121
- [Background] Warner MA, Meyerhoff KL, Warner ME, Posner KL, Stephens L, Domino KB. Pulmonary Aspiration of Gastric Contents: A Closed Claims Analysis. Anesthesiology. 2021 Aug 1;135(2):284-291. doi: 10.1097/ALN.0000000000003831. PMID 34019629
- [Background] Cook-Sather SD, Tulloch HV, Cnaan A, Nicolson SC, Cubina ML, Gallagher PR, Schreiner MS. A comparison of awake versus paralyzed tracheal intubation for infants with pyloric stenosis. Anesth Analg. 1998 May;86(5):945-51. doi: 10.1097/00000539-199805000-00006. PMID 9585274
- [Background] Evain JN, Durand Z, Dilworth K, Sintzel S, Courvoisier A, Mortamet G, Desgranges FP, Bouvet L, Payen JF. Assessing gastric contents in children before general anesthesia for acute extremity fracture: An ultrasound observational cohort study. J Clin Anesth. 2022 May;77:110598. doi: 10.1016/j.jclinane.2021.110598. Epub 2021 Nov 18. PMID 34801888
- [Background] Spencer AO, Walker AM, Yeung AK, Lardner DR, Yee K, Mulvey JM, Perlas A. Ultrasound assessment of gastric volume in the fasted pediatric patient undergoing upper gastrointestinal endoscopy: development of a predictive model using endoscopically suctioned volumes. Paediatr Anaesth. 2015 Mar;25(3):301-8. doi: 10.1111/pan.12581. Epub 2014 Dec 11. PMID 25495405
- [Background] Schmitz A, Schmidt AR, Buehler PK, Schraner T, Fruhauf M, Weiss M, Klaghofer R, Kellenberger CJ. Gastric ultrasound as a preoperative bedside test for residual gastric contents volume in children. Paediatr Anaesth. 2016 Dec;26(12):1157-1164. doi: 10.1111/pan.12993. Epub 2016 Aug 20. PMID 27543559
- [Background] Raidoo DM, Rocke DA, Brock-Utne JG, Marszalek A, Engelbrecht HE. Critical volume for pulmonary acid aspiration: reappraisal in a primate model. Br J Anaesth. 1990 Aug;65(2):248-50. doi: 10.1093/bja/65.2.248. PMID 2223347
- [Background] Cook-Sather SD, Liacouras CA, Previte JP, Markakis DA, Schreiner MS. Gastric fluid measurement by blind aspiration in paediatric patients: a gastroscopic evaluation. Can J Anaesth. 1997 Feb;44(2):168-72. doi: 10.1007/BF03013006. PMID 9043730
- [Result] Bricker SR, McLuckie A, Nightingale DA. Gastric aspirates after trauma in children. Anaesthesia. 1989 Sep;44(9):721-4. doi: 10.1111/j.1365-2044.1989.tb09255.x. PMID 2802116